CLINICAL TRIAL: NCT07202390
Title: Intraarticular Gold Microparticles for Knee Osteoarthritis. A Randomized Trial
Brief Title: Intraarticular Gold Microparticles for Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Sten Rasmussen, MD, PhD, Professor, Aalborg University Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GAIN XVI Knee RCT
Record Dates: First submitted 2025-09-05; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis
Keywords: Intraarticular gold; knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid; Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraarticular gold microprarticles plus hyaluronic acid (Experimental): 20 mg metallic gold microparticles (72.000 particles, 20-40 µm) will be injected into the knee joint using 2 mL hyaluronic acid.
  Interventions: Other: 20 mg metallic gold microparticles (72.000 particles, 20-40 µm) will be injected into the knee joint using 2 mL hyaluronic acid.; Other: Intervention
- Intraarticular hyaluronic acid (Placebo Comparator): 2 mL hyaluronic acid will be injected into the knee joint
  Interventions: Other: 20 mg metallic gold microparticles (72.000 particles, 20-40 µm) will be injected into the knee joint using 2 mL hyaluronic acid.; Other: Intervention

INTERVENTIONS:
Other: 20 mg metallic gold microparticles (72.000 particles, 20-40 µm) will be injected into the knee joint using 2 mL hyaluronic acid. — 20 mg metallic gold microparticles (72.000 particles, 20-40 µm) will be injected into the knee joint using 2 mL hyaluronic acid.
Other: Intervention — 20 mg metallic gold microparticles (72.000 particles, 20-40 µm) will be injected into the knee joint using 2 mL hyaluronic acid.

SUMMARY:
The investigators have shown in three pilot studies that intra-articular metallic gold microparticles can reduce knee osteoarthritis pain for up to two years. These results are noteworthy considering the growing number of older adults who suffer from osteoarthritis pain, which contributes to increased demand on healthcare resources. Demonstrating effective treatment could alleviate this burden for a significant portion of the aging population.

The specific aim is to evaluate whether intra-articular metallic gold microparticles are superior to placebo in reducing the need for additional treatment in patients with knee osteoarthritis within one year. The investigators will test the hypothesis that intra-articular metallic gold microparticles reduce subsequent treatment events by more than 50% compared to placebo during this period.

DETAILED DESCRIPTION:
To test the superiority of metallic gold microparticles over a placebo, 240 patients will be included in a randomized, double-blind, controlled trial. This process will take place over a period of 1-2 years. The study will follow the CONSORT Guidelines and comply with the Danish Data Protection Agency. The investigators will handle all data in an electronic form, including demographics and all outcome measures. The investigators will use an electronic Case Report Form (CRF). The management of data will be handled according to the Danish Data Protection Agency's guidelines. The host for data will be physically located at Aalborg University Research Data host, and at North Denmark Region, q-drive host, and follow the Guidelines from The Danish Protection Agency. The schedule for randomization will be randomly generated using a computer before the initiation of the trial. The medical doctor will be blind to group allocation and will not be involved in providing the metallic gold microparticles or placebo. The participants and the medical doctor performing follow-up will be blind to group allocation.

All patients will receive either intra-articular metallic gold microparticles and HA or HA alone. With the use of 2 cc syringe, the investigators will perform intra-articular injection using the standard approach for knee puncture and injection. For intervention, 20 mg metallic gold microparticles (72.000 particles, 20-40 µm) will be injected into the joint using 2 mL hyaluronic acid. For control, 2 mL of hyaluronic acid will be injected into the joint. A centralized computer-generated randomization will allocate to either 2 cc of hyaluronic acid with or without 20 mg metallic gold microparticles.

At the end of the trial, the patients in the control group will receive the intervention treatment with metallic gold microparticles.

ELIGIBILITY:
Inclusion Criteria:

* more than 6 months of knee pain without efficacy on pain of conservative treatment, radiographic knee osteoarthritis according to Kellgren-Lawrence grade 1-4, and age ≥18years

Exclusion Criteria:

* malalignment, indication for knee replacement surgery, malignancy, active infection and antibiotic treatment, active treatment with steroids, biological or other anti-Rheumatic medication, inability to comply with the protocol, inadequacy in the written and spoken national language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is any additional treatment event such as, re-referral, intra-articular injection, arthroscopy or any knee replacement surgery within 1 year. | 1 year
  Time to event

SECONDARY OUTCOMES:
The PainDetect questionnaire | 1 year
  The PainDetect questionnaire (Freynhagen et al., 2006) includes three components: gradation of pain, pain course pattern, and radiating pain. Gradation is measured by seven patient-scored questions on a 0 to 5 scale (0 = never; 5 = very strongly). Pain course pattern is assessed with one question where patients select one of four images, each representing a specific score (0, -1, or +1; two images may score +1). Radiating pain is determined by a yes (score +2) or no (score 0) response. Total scores span from -1 (no pain symptoms) to 38 (severe pain symptoms).
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 1 year
  The WOMAC questionnaire includes 24 questions: 5 for pain, 2 for stiffness, and 17 for physical function, each scored on a 5-point scale from 0 (none) to 4 (extreme). The summarized score span from 0 (no symptoms) to 96 (severe symptoms).
The quality of life score EQ-5D-5L | 1 yar
  The EQ-5D-5L (33) consists of two parts, a descriptive system and the EQ VAS. The descriptive system measures five dimensions of health: MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION. Each dimension has five response levels: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. For instance, 'slight problems' (e.g. 'I have slight problems in walking about') is always coded as '2'. The digits for the five dimensions can be combined in a 5-digit code that describes the respondent's health state profile; for instance, 21111 means slight problems in the mobility dimension and no problems in any of the other dimensions. The EQ VAS records the respondent's overall current health on a vertical visual analogue scale from 0 to 100, where "0" is "The best health you can imagine" and 100 "The worst health you can imagine
Proteomic analysis of synovial fluid and serum | 8 weeks
  The analyses of the proteomic primary raw data output from synovial fluid and serum obtained before and 8 weeks after treatment in both arms will be searched against spectral databases generated by fractionated pooled samples using human reference proteome database in Biognosys Spectronaut (Schaab et al., 2012) and using statistical analysis (Koh et al., 2019). Quantitative proteome analysis of synovial and serum samples will be accomplished by discovery proteomics using DIA-PASEF (Meier et al., 2020). Functional association of significantly regulated proteins in synovial fluid and serum with gene ontology and function will be asessed by Metascape.

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the study:
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: February 2029
URL: https://vbn.aau.dk/da/persons/sten

REFERENCES:
- [Background] Barfod KW, Blond L, Mikkelsen RK, Bagge J, Holmich LR, Kallemose T, Troelsen A, Holmich P. Treatment of knee osteoarthritis with a single injection of autologous micro-fragmented adipose tissue is not superior to a placebo saline injection: a blinded randomised controlled trial with 2-year follow-up. Br J Sports Med. 2025 Aug 26;59(17):1219-1227. doi: 10.1136/bjsports-2024-108732. PMID 40101939
- [Background] Kim KI, Kim MS, Kim JH. Intra-articular Injection of Autologous Adipose-Derived Stem Cells or Stromal Vascular Fractions: Are They Effective for Patients With Knee Osteoarthritis? A Systematic Review With Meta-analysis of Randomized Controlled Trials. Am J Sports Med. 2023 Mar;51(3):837-848. doi: 10.1177/03635465211053893. Epub 2022 Jan 12. PMID 35019764
- [Background] Peck J, Slovek A, Miro P, Vij N, Traube B, Lee C, Berger AA, Kassem H, Kaye AD, Sherman WF, Abd-Elsayed A. A Comprehensive Review of Viscosupplementation in Osteoarthritis of the Knee. Orthop Rev (Pavia). 2021 Jul 10;13(2):25549. doi: 10.52965/001c.25549. eCollection 2021. PMID 34745480
- [Background] Pereira TV, Juni P, Saadat P, Xing D, Yao L, Bobos P, Agarwal A, Hincapie CA, da Costa BR. Viscosupplementation for knee osteoarthritis: systematic review and meta-analysis. BMJ. 2022 Jul 6;378:e069722. doi: 10.1136/bmj-2022-069722. PMID 36333100
- [Background] Richard MJ, Driban JB, McAlindon TE. Pharmaceutical treatment of osteoarthritis. Osteoarthritis Cartilage. 2023 Apr;31(4):458-466. doi: 10.1016/j.joca.2022.11.005. Epub 2022 Nov 19. PMID 36414224
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] Altman RD, Devji T, Bhandari M, Fierlinger A, Niazi F, Christensen R. Clinical benefit of intra-articular saline as a comparator in clinical trials of knee osteoarthritis treatments: A systematic review and meta-analysis of randomized trials. Semin Arthritis Rheum. 2016 Oct;46(2):151-159. doi: 10.1016/j.semarthrit.2016.04.003. Epub 2016 Apr 27. PMID 27238876
- [Background] Patel S, Dhillon MS, Aggarwal S, Marwaha N, Jain A. Treatment with platelet-rich plasma is more effective than placebo for knee osteoarthritis: a prospective, double-blind, randomized trial. Am J Sports Med. 2013 Feb;41(2):356-64. doi: 10.1177/0363546512471299. Epub 2013 Jan 8. PMID 23299850
- [Background] Bellamy N, Campbell J, Robinson V, Gee T, Bourne R, Wells G. Intraarticular corticosteroid for treatment of osteoarthritis of the knee. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD005328. doi: 10.1002/14651858.CD005328.pub2. PMID 16625636
- [Background] Chavda S, Rabbani SA, Wadhwa T. Role and Effectiveness of Intra-articular Injection of Hyaluronic Acid in the Treatment of Knee Osteoarthritis: A Systematic Review. Cureus. 2022 Apr 26;14(4):e24503. doi: 10.7759/cureus.24503. eCollection 2022 Apr. PMID 35651409
- [Background] Bhandari M, Bannuru RR, Babins EM, Martel-Pelletier J, Khan M, Raynauld JP, Frankovich R, Mcleod D, Devji T, Phillips M, Schemitsch EH, Pelletier JP. Intra-articular hyaluronic acid in the treatment of knee osteoarthritis: a Canadian evidence-based perspective. Ther Adv Musculoskelet Dis. 2017 Sep;9(9):231-246. doi: 10.1177/1759720X17729641. Epub 2017 Sep 12. PMID 28932293
- [Background] Concoff A, Sancheti P, Niazi F, Shaw P, Rosen J. The efficacy of multiple versus single hyaluronic acid injections: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2017 Dec 21;18(1):542. doi: 10.1186/s12891-017-1897-2. PMID 29268731
- [Background] Skou ST, Rasmussen S, Laursen MB, Rathleff MS, Arendt-Nielsen L, Simonsen O, Roos EM. The efficacy of 12 weeks non-surgical treatment for patients not eligible for total knee replacement: a randomized controlled trial with 1-year follow-up. Osteoarthritis Cartilage. 2015 Sep;23(9):1465-75. doi: 10.1016/j.joca.2015.04.021. Epub 2015 Apr 30. PMID 25937024
- [Background] Skou ST, Roos EM, Laursen MB, Rathleff MS, Arendt-Nielsen L, Simonsen O, Rasmussen S. A Randomized, Controlled Trial of Total Knee Replacement. N Engl J Med. 2015 Oct 22;373(17):1597-606. doi: 10.1056/NEJMoa1505467. PMID 26488691
- [Background] Zhang Z, Hu Z, Zhao D, Huang H, Liang Y, Mao B. Arthroscopic surgery is not superior to conservative treatment in knee osteoarthritis: a systematic review and meta-analysis of randomized controlled trails. BMC Musculoskelet Disord. 2024 Sep 5;25(1):712. doi: 10.1186/s12891-024-07813-3. PMID 39237972
- [Background] Cotter EJ, Weissman AC, Yazdi AA, Muth SA, Cole BJ. Arthroscopic Debridement of Mild and Moderate Knee Osteoarthritis Results in Clinical Improvement at Short-Term Follow-Up: A Systematic Review. Arthroscopy. 2025 Feb;41(2):377-389. doi: 10.1016/j.arthro.2024.03.016. Epub 2024 Mar 18. PMID 38508289
- [Background] Petterson SC, Brite JE, Jelen ES, Wang KH, Reyes MM, Briggs KK, Plancher KD. Arthroscopic Management of Moderate-to-Severe Osteoarthritis of the Knee: A Systematic Review. JBJS Rev. 2024 Sep 19;12(9). doi: 10.2106/JBJS.RVW.24.00100. eCollection 2024 Sep 1. PMID 39348469
- [Background] Turkiewicz A, Gerhardsson de Verdier M, Engstrom G, Nilsson PM, Mellstrom C, Lohmander LS, Englund M. Prevalence of knee pain and knee OA in southern Sweden and the proportion that seeks medical care. Rheumatology (Oxford). 2015 May;54(5):827-35. doi: 10.1093/rheumatology/keu409. Epub 2014 Oct 13. PMID 25313145
- [Background] Cao F, Xu Z, Li XX, Fu ZY, Han RY, Zhang JL, Wang P, Hou S, Pan HF. Trends and cross-country inequalities in the global burden of osteoarthritis, 1990-2019: A population-based study. Ageing Res Rev. 2024 Aug;99:102382. doi: 10.1016/j.arr.2024.102382. Epub 2024 Jun 23. PMID 38917934
- [Background] Li XX, Cao F, Zhao CN, Ge M, Wei HF, Tang J, Xu WL, Wang S, Gao M, Wang P, Pan HF. Global burden of osteoarthritis: Prevalence and temporal trends from 1990 to 2019. Int J Rheum Dis. 2024 Aug;27(8):e15285. doi: 10.1111/1756-185X.15285. PMID 39114972
- [Background] Rasmussen S, Skjoldemose E, Jorgensen NK. Intraarticular gold microparticles using hyaluronic acid as the carrier for hip osteoarthritis. A 2-year follow-up pilot study. Sci Rep. 2024 Nov 1;14(1):26249. doi: 10.1038/s41598-024-77760-5. PMID 39482349
- [Background] Rasmussen S, Aboo C, Skallerup J, Stensballe A. Intraarticular gold for knee osteoarthritis: An ancillary analysis of biomarkers and outcome of a pilot study. Osteoarthr Cartil Open. 2024 Aug 31;6(4):100514. doi: 10.1016/j.ocarto.2024.100514. eCollection 2024 Dec. PMID 39291082
- [Background] Rasmussen S, Frederickson C, Danscher G. Inhibition of Local Inflammation by Implanted Gold: A Narrative Review of the History and Use of Gold. J Rheumatol. 2023 May;50(5):704-705. doi: 10.3899/jrheum.221150. Epub 2023 Mar 15. No abstract available. PMID 36921973
- [Background] Danscher G, Rasmussen S. nanoGold and microGold inhibit autoimmune inflammation: a review. Histochem Cell Biol. 2023 Mar;159(3):225-232. doi: 10.1007/s00418-023-02182-9. Epub 2023 Mar 2. PMID 36864314
- [Background] Rasmussen S, Kjaer Petersen K, Kristiansen MK, Skallerup J, Aboo C, Thomsen ME, Skjoldemose E, Jorgensen NK, Stensballe A, Arendt-Nielsen L. Gold micro-particles for knee osteoarthritis. Eur J Pain. 2022 Apr;26(4):811-824. doi: 10.1002/ejp.1909. Epub 2022 Feb 1. PMID 35076138